CLINICAL TRIAL: NCT02327910
Title: The Clinical Value of Applying Qualitative TOF Monitoring and Transcutaneous Partial Pressure of Carbon Dioxide to Guide Elderly Patients Extubation
Brief Title: The Clinical Value of Applying TOF and TcPO2 to Guide Elderly Patients Extubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Zhaolei, The medical team leader, Beijing Municipal Science & Technology Commission
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BeijingMSTC
Record Dates: First submitted 2014-12-20; First posted 2014-12-31 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2015-12

CONDITIONS: Postoperative Respiratory Complications
Keywords: Elderly patients，; General anesthesia，; Transcutaneous partial pressure of carbon dioxide(TcPCO2)，; Train-of-four(TOF)，; Extubation; ，Respiratory events

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conventional group (No Intervention): Conventional group:The patients of conventional group were extubated when standard criteria were met;
- TOF group (Experimental): TOF group: patients had a TOF ratio of greater than 0.90 as an additional extubation criterion;
  Interventions: Other: TOF group
- TOF unit TcPCO2 group (Experimental): Qualitative TOF and transcutaneous partial pressure of carbon dioxide monitoring(Unite group):the patients of U group were extubated when TOF ratio greater than 0.9 and TcPCO2 recovery to preoprative(±5mmHg)
  Interventions: Other: TOF unit TcPCO2 group

INTERVENTIONS:
Other: TOF unit TcPCO2 group — The patients of U group were extubated when TOF ratio greater than 0.9 and TcPCO2 recovery to preoprative(±5mmHg)
  Arms: TOF unit TcPCO2 group
Other: TOF group — The patients of T group were extubated when TOF ratio greater than 0.9.
  Arms: TOF group

SUMMARY:
Three hundred aged(age>65y) patients were randomized to Commom group(C group). Qualitative TOF monitoring (TOF group). Qualitative TOF and transcutaneous partial pressure of carbon dioxide monitoring(Unite group). Anesthetic management was standardized in all subjects .The patients of C group were extubated when standard criteria were met; T group patients had a TOF ratio of greater than 0.90 as an additional extubation criterion;and U group patiens were extubated when TOF ratio is greater than 0.90 and meanwhile transcutaneous partial pressure of carbon dioxide recovered to preoperative ±5mmHg .All the patients were transport to the PACU after extubation.Compare the adverse respiratory events at the moment of extubation, on the arrival of PACU, at 30min and 60min moment in the PACU respectively.

DETAILED DESCRIPTION:
Three hundred aged(age>65y) patients were rondomized to acceleromyographic monitoring unit transcutaneous CO2 partial pressure(TcPCO2) monitoring(U group)or acceleromyographic monitering(T group)or conventional(C group).Anesthethic management was standardized.U patients were extubated when TOF ratio greater than 0.9 and transcutaneous CO2 partial pressure recover to preoprative (±5mmHg).T patients were extubated when TOF ratio greater than 0.9.C patients were extubated when standard criteria were met.Anesthesia monitoring, including ECG, invasive arterial pressure, pulse oxygen saturation, the BIS, nasopharyngeal temperature.The anesthesia induction with propofol 1 ~ 2 mg/kg, rocuronium 0.6 mg/kg, fentanyl 2 ug/kg, anesthesia maintained using propofol, fentanyl and the rocuronium 0.3 mg/kg. continuous pumping, maintain circulation stabilization and BIS value in 40 ~ 60, about 30 minutes before the end of surgery to stop rocuronium infusion, at the end of sewing leather to stop propofol and fentanyl infusion. Adjust Respiratory parameters, maintain breathe out co2 partial pressure at the scope of the 30 ~ 35 MMHG, using the variable temperature blanket insulation. All patients are monitored and give the muscle relaxant antagonists, pulling out endotracheal intubation, recording the TOF and TcPCO2 data when leaving the operating room . But during anesthesia management in group C, shielding TOF and TcPCO2 data to the anesthesiologists; T group during anesthesia management, shielding TcPCO2 data to the anesthesiologist; U set during anesthesia management, can according to the TOF and TcPCO2 data to management. All postoperative patients are sent into PACU, giving oxygen mask 3L/min, they can leave PACU Aldrete score nine points or more. By blind method principle, physicians of PACU,who is responsible for the patients with postoperative index records and statistics are blind to the staff for grouping, intraoperative management and BiBa tube drawing situation , in order to avoid bias. Statistical analysis: all the data represented as mean + / - standard deviation, using SPSS statistical software, measuring data comparison using analysis of variance between groups, count data using chi-square test, P < 0.05 that was statistically significant

ELIGIBILITY:
Inclusion Criteria:

* Elective general anesthesia surgery elderly patients (age > 65 years), gastrointestinal surgery

Exclusion Criteria:

* ASA grade III or IV level, merging, bronchial asthma, chronic obstructive pulmonary disease, severe liver and kidney function is not complete (liver and kidney function corresponding biochemical index 50% above the normal level), neuromuscular disease, and use effect of neuromuscular transmission drugs or severe obesity (BMI > 35) of the patients

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
The comparison between groups of postoperative respiratory adverse events | up to 24 month

IPD SHARING:
Plan to Share IPD: Yes